CLINICAL TRIAL: NCT02690805
Title: Predicting Neoadjuvant Chemotherapy Response by Using a Combined MRI and Scinti-Mammography (MRI-SMM) System
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: UCI HS# 2015-1866
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients receiving neoadjuvant chemotherapy: One arm: Combined MRI-SMM Imaging
  Interventions: Device: MR-compatible scinti-mammography (MRI-SMM) system

INTERVENTIONS:
Device: MR-compatible scinti-mammography (MRI-SMM) system

SUMMARY:
The purpose of this research study is to investigate the accuracy of a breast imaging system that measures the uptake of the injected radioactive tracer by gamma-ray imaging, known as scinti-mammography (SMM), to diagnose the residual breast cancer after neoadjuvant chemotherapy (NAC) treatment by comparing to MRI.

DETAILED DESCRIPTION:
The optimal goal of neoadjuvant chemotherapy (NAC) for breast cancer is to achieve pathologic complete response (pCR) with the least toxicity. As more effective therapies become available, one challenge is how to evaluate the response of tumor in a timely manner, so an optimal regimen can be given to the patient. Reliable imaging methods that can monitor and predict NAC response are needed. MRI is known as the most accurate imaging modality to evaluate the response to NAC based on tumor shrinkage, but so far there is no reliable parameter that can be measured at early times after the administration of drugs to predict the final treatment outcome. Furthermore, some patients may have contradiction to receive MRI, or cannot tolerate the long scan time in a prone position. Other imaging modalities that can measure early functional (particularly metabolic) changes are being investigated, and have shown some success. In this study investigators will assess the role of an MR-compatible scinti-mammography (MRI-SMM) system for monitoring and predicting NAC response. A total of 75 breast cancer patients receiving NAC will be enrolled, and each subject will receive 3 imaging studies before, during, and after completing NAC. The aims are: 1) to compare the tumor size measured by SMM and MRI at different times; 2) to evaluate the respective diagnostic accuracy of the post-NAC residual disease measured by SMM and MRI by comparing to pathological examination results as the gold standard; 3) to investigate the respective and combined ability of MRI and SMM, based on pre-treatment and early changes in the first follow-up imaging, for predicting pathologic complete response (pCR). The diagnostic results obtained using MRI and SMM from tumors of varying stages at different times during NAC will provide important information for establishing the role of a standalone SMM system, as well as the combined MRI-SMM system, for management of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. A female older than 21 years of age,
2. Have biopsy-proven breast cancer and decided to receive neoadjuvant chemotherapy.
3. Are in good health (other than having breast cancer) and can lie still in a prone position for 45 minutes inside MRI scanner.

Exclusion Criteria:

1. Pregnant,
2. Unwilling to give informed consent,
3. Have implanted prosthetic heart valves, pacemaker, neuro-stimulation devices, surgical clips (hemostatic clips) or other metallic implants,
4. Have engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials (e.g. iron), or have imbedded metal fragments from military activities,
5. Have received orthodontic work involving ferromagnetic materials,
6. Claustrophobic (i.e. feeling very anxious in a confined small space),
7. Have had allergic response to contrast agents (such as iodine or gadolinium) previously,
8. Have known history of kidney diseases.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who elect to receive neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of residual breast cancer after neoadjuvant chemotherapy as assessed by MRI and scinti-mammography | 3 years
  Breast cancer patients receiving neoadjuvant chemotherapy will be imaged by a combined MRI and scinti-mammography (MRI-SMM) imaging system, and the diagnostic accuracy as assessed by MRI and SMM will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No